CLINICAL TRIAL: NCT03920657
Title: Early and Low Dose Deferasirox (3.5 mg/kg FCT) to Suppress NTBI and LPI as Early Intervention to Prevent Tissue Iron Overload in Lower Risk MDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment failed
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FISM_IRON-MDS
Record Dates: First submitted 2018-12-14; First posted 2019-04-19 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2021-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Deferasirox

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm, phase II, study designed to look whether early intervention with low dose DFX improves clinical outcome of patients with MDS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferasirox (Experimental): patients will be assigned to a fixed dose of 3.5 mg/kg/day of DFX FCT.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Fixed dose of 3.5 mg/kg/day of DFX FCT
  Other Names: Exjade

SUMMARY:
The scientific rationale for this study is the evolving understanding that iron-induced tissue damage is not only a process of progressive bulking of organs through high-volumes iron deposition, but also a reactive iron species related "toxic" damage.

Iron mediated damage can occur prior reaching high iron storage thresholds derived from thalassemia major setting, free toxic iron species being already present when transferrin saturation >60-70% (25); therefore a timely early adoption of iron chelation may be of benefit before overt iron overload is seen.

Our hypothesis is that early and low dose DFX-FCT is better tolerated and is able to prevent iron accumulation and consequently tissue iron related damage, by consistently suppressing iron reactive oxygen species (NTBI and LPI).

If this hypothesis is confirmed this approach could contribute to an improvement of clinical practice of patients managements. Additionally this approach might also be a contribute in preventing future iron overloaded related complication, in this already frail and co-treated patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Adult Myelodysplastic Syndrome (≥18 years).
* Revised IPSS: very low. low - intermediate
* Having received 5-20 packed red blood cell units
* Serum ferritin ≥300 ng/ml
* Transferrin saturation ≥ 60%
* Chelation naïve
* Capability to provide informed consent

Exclusion Criteria:

* Patients aged <18 years old
* Higher risk (revised IPSS) MDS (Intermediate 2, high)
* Cumulative transfusion story of > 20 packed red cell units
* Creatinine Clearance (CrCL): <60 ml/min. Patients with CrCl of 40-60ml/min will be included only individually if no other renal risk factors are present.
* Serum creatinine >2 x ULN at screening. If borderline serum creatinine will be measured within 7-10 days and the mean value will be used for eligibility criteria.
* Significant proteinuria as indicated by a urinary protein/creatinine ratio > 0.5 mg/mg in a non-first void urine sample (or alternatively in two of three samples obtained for screening).
* ECOG performance status >2.
* Left ventricular ejection fraction < 50% by echocardiography
* A history of repeated hospitalization for congestive heart failure.
* Systemic diseases that would prevent study treatment (e.g. uncontrolled hypertension, cardiovascular, renal, hepatic, metabolic, etc.)
* Clinical or laboratory evidence of chronic Hepatitis B or Hepatitis C (definition of chronic hepatitis follows EASL 2017 criteria).
* History of HIV positive test result (ELISA or Western blot).
* Treatment with systemic investigational drug within 4 weeks or topical investigational drug within 7 days of study start.
* ALT or AST over 3 times superior to ULN at screening.
* ANC < 500/ microL
* Platelets transfusion dependency
* Total bilirubin over 1.5 times superior to ULN at screening (patients with Gilbert syndrome are allowed to enter the study)
* Diagnosis of Child score C liver cirrhosis.
* Patients participating in another clinical trial other than an observational registry study.
* Patients with a history of another malignancy within the past 3 years, with the exception of basal skin carcinoma or cervical carcinoma in situ or completely resected colonic polyps carcinoma in situ.
* History of non-compliance to medical regimens, or patients who are considered potentially unreliable and/or not cooperative.
* Presence of a surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug.
* Pregnant, intending-to-become pregnant, or breast-feeding patients.
* Women of potential maternity age who do not agree to practice effective contraceptive methods fo the entire study duration.
* History of drug or alcohol abuse within the 12 months prior to enrollment.
* Hypersensitivity to the active substance or to any of the excipients.
* Inability to provide a valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Change of hepatic iron | 1 year
  Change of hepatic iron from the baseline according to baseline hepatic iron level: For patients with baseline LIC ≤5 mg/g dry weight (dw) ± 1.5 mg/g dw. For patients with baseline LIC >5 mg/g dw ±20%

SECONDARY OUTCOMES:
Definition of iron overload | 1 year
  The baseline iron status of MDS patients at the beginning of their transfusion story is today unknown. This study is the first unbiased and direct measurement of iron stress and oxidative stress in MDS patients at the beginning of the transfusion story.
  Baseline iron status will be described by classical iron markers:
  serum ferritin (ng/ml), transferritin saturation (%), liver and pancreas iron concentration by MRI (mg/g dry weight). Total body iron stores will be calculated (mg/kg) with the published formula (N Engl J Med 2000; 343:327-331).
  Tissue reactive oxygen species will be measured in the patient's plasma as follows:
  non-transferrin bound iron= micromoles/L, Labile Plasma Iron= micromoles/L. Oxidative stress will be measured by Malonildialdehyde (MDA). Levels in plasmas= micromoles/L.
Efficacy of treatment | 1 year
  Absolute change in hepatic iron concentration EOS versus baseline.
Evolution of iron overload serologic markers | 1 year
  Absolute and relative changes in serum ferritin and transferrin saturation from baseline to every visit during the whole treatment period
Evolution of toxic serum iron forms | 1 year
  Presence and quantitative evolution of toxic serum iron forms (iron tissue reactive species) under low dose DFX therapy
Relationship between NTBI and LPI with serum ferritin and liver and pancreas iron overload | 1 year
  Prevention of iron overload will be studied by the difference iron parameters end of therapy - baseline by liver iron concentration (mg/g dry weight), pancreas iron concentration (mg/g dry weight), total body iron stores (mg/kg) calculated the N Engl J med 2000 343:327-331 formula = liver iron concentration x 10.6.
  Serum ferritin = ng/ml.
  Relationship between suppression of tissue iron species and prevention of iron accumulation (observational study) will be measured by the:
  NTBI/LPI values (micromoles/L), Differences end of study - baseline quantitative parameters of iron loading (liver and pancreas iron concentration and total body iron stores).
Overall safety of deferasirox | 1 year
  Evaluate the overall safety of deferasirox FCT formulation in patients with lower risk MDS at the beginning of their transfusional history
Leukemic transformation | 1 year
  Leukemic transformation (progression to leukemia or higher rIPSS scores)
Hemopoietic response | 1 year
  Percentage of patients with hematologic improvements in term of erythroid response following IWG 2006 criteria.
Costs analysis | 1 year
  Treatment cost will be compared with standard approach cost (14 mg/kg/day. DFX-FCT after 20 units of packed red cells units and serum ferritin> 1000 ng/ml over one year of treatment). For comparison literature and matched FISM registry data will be used. Unit of measurement will be 2019 USD and Euros.
Study of biological cellular damage | 1 year
  Biological cellular damage will be measured by presence and level of oxidative stress determined at baseline, during and at end of study and compared with ongoing treatment by: Malonildialdehyde (MDA) plasma levels (micromoles/L).

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - S.O.D. Ematologia Policlino Careggi, Florence, FI
  - Medicina Interna II Divisione di Ematologia, Ospedale S. Luigi Gonzaga, Orbassano, TO
  - Ematologia - Spedali Civili, Brescia
  - Ospedale Businco, Cagliari
  - Ospedale San Martino, Genova
  - Ospedale Niguarda, Milan
  - Azienda Ospedaliera di Padova, Padua
  - AO Bianchi Melacrino Morelli, Reggio Calabria
  - Ospedale S. Eugenio, Roma
  - Istituto clinico Humanitas, Rozzano (MI)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03920657/Prot_SAP_000.pdf